CLINICAL TRIAL: NCT04051762
Title: A Comparative Study Between Postextubation of Preterm Infants Into High-Flow Nasal Cannulae V.S Nasal Continuous Positive Airway Pressure
Status: Completed | Type: Observational
Sponsor: Ramy Saleh Morsy (Other)
Responsible Party: Sponsor-Investigator, Ramy Saleh Morsy, Assistatnt Lecturer in AFCM, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Post extubation HFNC vs. NCPAP
Record Dates: First submitted 2019-07-03; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm neonates on HFNC: neonates extubated to HFNC (High flow nasal cannula)
  Interventions: Device: High flow nasal cannula vs. Nasal continuous positive airway pressure
- Preterm neonates on NCPAP: neonates extubated to NCPAP ( nasal continuous positive airway pressure)
  Interventions: Device: High flow nasal cannula vs. Nasal continuous positive airway pressure

INTERVENTIONS:
Device: High flow nasal cannula vs. Nasal continuous positive airway pressure — High flow nasal cannula

SUMMARY:
The investigators hypothesize that there is a growing trend of the feasibility of HFNC as an alternative to other forms of non-invasive ventilation mechanism to provide continuous distending pressure to preterm infants. However, there remains uncertainty about the efficacy and safety of HFNC in this population.

DETAILED DESCRIPTION:
Our primary outcome is to determine whether postextubation respiratory support via heated humidified high-flow nasal cannula results in a greater proportion of infants younger than 34 weeks gestation being successfully extubated after a period of endotracheal positive pressure ventilation compared with conventional (NCPAP).

The following study will be conducted in the neonatal intensive care unit (NICU) of Gynecology and Obstetric department of Kasr El Aini hospital and neonatal intensive care unit of Military Hospital throughout a time interval of at least 6 months for a minimum of 100 preterm infants.

Infants will be eligible for the study if they born at less than 34 weeks' gestation, required endotracheal intubation and positive pressure ventilation, and considered ready for extubation by the clinical team.

The investigators will assign extubation of preterm ventilated infants (50 preterm infant) in NICU of Military Hospital into HHFNC and extubation of preterm ventilated infants (50 preterm infant) in (NICU) of Gynecology and Obstetric department of Kasr El Aini hospital into NCPAP (50 preterm infant).

ELIGIBILITY:
Inclusion Criteria:

•Infants born at a gestational age of less than 34 weeks, receiving mechanical ventilation through an endotracheal tube.

Exclusion Criteria:

* Full term neonates or large for gestational age.
* Preterm neonates not supported primarily by invasive ventilation.
* Infants with suspected upper airway obstruction, congenital airway malformations or major cardiopulmonary malformations.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The following study will be conducted in the neonatal intensive care unit (NICU) of Gynecology and Obstetric department of Kasr El Aini hospital and neonatal intensive care unit of Military Hospital throughout a time interval of at least 6 months for a minimum of 100 preterm infants.
  Infants will be eligible for the study if they born at less than 34 weeks' gestation, required endotracheal intubation and positive pressure ventilation, and considered ready for extubation by the clinical team.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
postextubation respiratory support | through study completion, an average of 1 year
  compare successful extubation of preterm (less than 34 weeks) into high flow nasal cannula versus continues positive airway pressure.

SECONDARY OUTCOMES:
postextubation respiratory support follow up | through study completion, an average of 1 year
  Secondary outcomes include the following:
  1. Need for delayed reintubation (beyond 7 days)
  2. Incidence of bronchopulmonary dysplasia.
  3. Total number of days of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Magda Mahmoud Badawy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No